CLINICAL TRIAL: NCT05244980
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group, Multi-Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TDM-105795 in Healthy Male Subjects With Androgenetic Alopecia (AGA)
Brief Title: A Study of TDM-105795 in Male Subjects With Androgenetic Alopecia (AGA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Technoderma Medicines Inc. (Industry)
Collaborators: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 239-11651-102
Record Dates: First submitted 2022-01-13; First posted 2022-02-17 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Alopecia, Androgenetic
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group, Multi-Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TDM-105795 in Healthy Male Subjects with Androgenetic Alopecia
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAD Cohorts 1-4 TDM-105795 topical solution (Experimental): Multiple dose administration of TDM-105795 Topical Solution, 0.0025% or 0.005% or 0.01% or 0.02%
  Interventions: Drug: TDM-105795
- Placebo for TDM-105795 topical solution (Placebo Comparator): Multiple dose administration of Placebo forTDM-105795 Topical Solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TDM-105795 — TDM-105795 topical solution
  Arms: MAD Cohorts 1-4 TDM-105795 topical solution
Drug: Placebo — Placebo for TDM-105795 topical solution
  Arms: Placebo for TDM-105795 topical solution

SUMMARY:
Multi-center, randomized, double-blind, vehicle-controlled, parallel group, multi-dose escalation study of TDM-105795 in male subjects, 18 to 55 years old, with Androgenetic Alopecia (AGA).

DETAILED DESCRIPTION:
Protocol 239-11651-102 is a planned Phase 1 study entitled "A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group, Multi-Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TDM-105795 in Healthy Male Subjects with Androgenetic Alopecia". Eligible subjects will be assigned to a sequential treatment cohort and will receive either one of the TDM-105795 solutions or the Placebo. The assigned test article will be applied once daily onto the scalp in the hair loss area (e.g., top of head and temple areas). All subjects will be treated with 1 mL/dose of test article with application to the scalp focusing on the regions that are bald and thinning.

ELIGIBILITY:
Inclusion Criteria:

To enter the study, a subject must meet the following criteria:

1. Subject is male, 18-55 years old.
2. Subject has provided written informed consent.
3. Subject has a clinical diagnosis of moderate to severe AGA in temple and vertex region, III to VI on the Modified Norwood-Hamilton Scale (i.e., III, IV, V, and VI).
4. Subject is willing and able to apply the test article(s) as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
5. Subject, in the investigator's opinion, is in good general health and free of any disease state or physical condition that might impair evaluation of AGA or exposes the subject to an unacceptable risk by study participation.
6. Subject has normal renal, thyroid, and hepatic function as determined by the Visit 1/Screening laboratory results in the opinion of the investigator.
7. Subject is a non-smoker, defined as not having smoked or used any form of tobacco or non-tobacco products containing nicotine in more than 6 months before Visit 2/Baseline.
8. Subject has a body mass index (BMI) of 19 to 32 kg/m2 inclusive and body weight not less than 50 kg at Visit 1/Screening.
9. Subject agrees to continue his other general hair care products and regimen for at least 2 weeks prior to Visit 2/Baseline, and through the entire study.
10. Subjects who are sexually active with a female partner and are not surgically sterile (vasectomy performed at least 6 months prior to treatment) must agree to refrain from sperm donation for at least 90 days after administration of their last dose of test article(s) and inform their non-pregant female sexual partner to use a highly effective form of birth control as described in the informed consent form. Note: Female partner must be confirmed according to subject to be non-pregnant at Visit 1/Screening and Visit 2/Baseline or at the visit when a subject identifies a new sexual partner.

Exclusion Criteria:

A subject is ineligible to enter the study if he meets 1 or more of the following criteria:

1. Subject has any dermatological disorders of the scalp on the regions that are bald and thinning with the possibility of interfering with the application of the test article or examination method, such as fungal or bacterial infections, seborrheic dermatitis, psoriasis, eczema, folliculitis, scars, or scalp atrophy.
2. Subject has any skin pathology or condition (e.g., uncontrolled thyroid disease, certain genetic disorders that involve hair growth or patterns) that, in the investigator's opinion, could interfere with the evaluation of the test article or requires use of interfering topical, systemic, or surgical therapy.
3. Subject has any visible inflammatory skin disease, injury, or condition of their scalp that could compromise subject safety and/or interfere with the evaluation of local or systemic assessments performed during the study.
4. Subject has a history of scalp reduction or notable trauma with related scarring, hair transplants, and/or hair weaves.
5. Subject has a known or suspected malignancy.
6. Subject has a positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody.
7. Subject has any condition, which, in the investigator's opinion, would make it unsafe for the subject to participate in this study, including clinically significant abnormal laboratory or 12-lead electrocardiogram (ECG) findings during the screening period or Visit 2/Baseline prior to dosing of the test article.
8. Subject has a hospital admission or major surgery within 30 days prior to Visit 2/ Baseline or planned for during the study.
9. Subject is currently enrolled in an investigational drug, biologic, or device study.
10. Subject has used an investigational drug, investigational biologic, or investigational device treatment within 30 days or 5 half-lives, whichever is longer, prior to Visit 2/Baseline.
11. Subject has a history of prescription drug abuse, or illicit drug use within 6 months prior to Visit 1/Screening.
12. Subject has a history of alcohol abuse according to medical history within 6 months prior to Visit 1/Screening.
13. Subject has a positive screen for alcohol or drugs of abuse at Visit 1/Screening or Visit 2/Baseline.
14. Subject has a donation or blood collection of more than 1 unit (approximately 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to Visit 2/Baseline.
15. A. Subject has used systemic inhibitors or inducers of CYP3A4 and Pgp (including rifampicin, rifabutin, St. John's Wort, corticosteroids, and environmental exposure) within 30 days prior to dosing at Visit 2/Baseline. B. Subject drank grapefruit juice within 7 days prior to dosing at Visit 2/Baseline.
16. Subject has used systemic prescription medications, herbals (including herbal teas and garlic extracts) supplements within 14 days prior to dosing at Visit 2/Baseline.
17. Subject has used systemic over the counter (OTC) medications or vitamins within 7 days prior to dosing at Visit 2/Baseline. (Note: Use of acetaminophen at < 3g/day is permitted until 24 hours prior to dosing at Visit 2/Baseline).
18. Subject has used any scalp hair growth treatments including medical devices (e.g., LED caps/wands/combs), prescription products (e.g., minoxidil, finasteride, dutasteride, etc.), herbal, homeopathy or other forms of treatment which may affect hair growth (in the opinion of the investigator) within 14 days prior to dosing at Visit 2/Baseline.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Incidence rate of any local and systemic AEs | 42 days
  Collection of adverse events
Number of subjects with presence (and severity) of local skin reactions (LSRs) | 42 days
  Collection of LSRs
Number of participants with abnormal vital signs | 28 days
  Collection of vital signs on day 1, day 8, and day 28
Number of participants with abnormal laboratory test results | 28 days
  Collection of safety labs at day 1, 8, 15, and 28
Number of participants with abnormal ECG readings | 28 days
  Collection of ECGs at day 1, 8, and 28
Number of participants with abnormal echocardiogram results | 38 days
  Collection of quantitative echo parameters at screening and EOT

SECONDARY OUTCOMES:
Plasma concentrations of TDM-105795 | 29 days
  Plasma concentrations of TDM-105795

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Piacquadio, M.D., Study Director — Therapeutics Incorporated
Locations (2):
- United States (2):
  - TCR Medical Corporation, San Diego, California
  - J&S Studies, Inc., College Station, Texas

IPD SHARING:
Plan to Share IPD: No